CLINICAL TRIAL: NCT05943054
Title: Role of the Striatum and Hippocampus on Different Time Scales
Brief Title: Striatum and Hippocampus on Different Time Scales
Acronym: e-Time
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP20211105; 2021-A01008-33 (Other: N° IDRCB)
Record Dates: First submitted 2022-03-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Huntington Disease; Alzheimer Disease
Keywords: Time processing; Huntington's disease; Alzheimer's disease; Striatum; Hippocampus
MeSH Terms: conditions — Huntington Disease; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients carrying the Huntington's gene (Experimental): A "long" temporal perception task and a "short" temporal perception task
  Interventions: Other: Temporal perception tasks
- Alzheimer's disease patients (Experimental): A "long" temporal perception task and a "short" temporal perception task
  Interventions: Other: Temporal perception tasks
- Healthy Volunteers (Active Comparator): A "long" temporal perception task and a "short" temporal perception task
  Interventions: Other: Temporal perception tasks

INTERVENTIONS:
Other: Temporal perception tasks — A "long" temporal perception task in which the duration of the stimulus, around 2 min, is materialized by a video. For each trial, two videos are displayed to the participants, and then the task of the participant is to indicate the longest video and to give his level of confidence in his answer. A "short" temporal perception task which will take place in the same way as the "long" task except that the duration of the stimulus, around 2 seconds, is materialized by still frames from the videos used in the previous task.

SUMMARY:
Time processing is fundamental to survival and goal reaching in humans. Different time scales (seconds, minutes, and beyond) are processed through specific cognitive processes involving different neural representations. It is generally agreed that time scale in seconds-to-minutes range named "interval timing" would be anatomically linked to the striatum. Indeed, it is possible to demonstrate a deficit of interval timing processes in patients suffering from striatal damage (Huntington's disease). However, recent findings show involvement of a second brain structure, the hippocampus, in interval timing processing in the minutes range, suggesting an interaction between the striatum and hippocampus. Presumably, patients with hippocampal damage (Alzheimer's disease) would specifically show a decrease in performance for this minutes-range time scale. This study aims to provide a better understanding of the role of the striatum in the treatment of time and its interactions with other brain structures such as the hippocampus. More specifically, it is unclear whether the striatum plays a platform role that would always be involved regardless of the time scale, as suggested by the unified model of time or whether different brain structures is solicited according to the time scale, as suggested by the modular system model. In order to elucidate these issues, a potential double dissociation between brain structures and time scales will be tested.

DETAILED DESCRIPTION:
In that aim, we will evaluate patients with Huntington's disease and patients with Alzheimer's disease by developing and using time processing paradigms comparing short and long time scales.

ELIGIBILITY:
Inclusion Criteria:

* Huntington's disease gene carriers

  * Patient included in the BioHD protocol
  * Age from 18 to 90 years old
  * Symptomatic patient
  * TFC ≥ 11
  * UHDRS motor> 5
  * Native language: French
  * Affiliation to a social security or to another social protection
  * Signature of informed consent

    • Patients with Alzheimer's disease
  * MMS from 20 to 26 (included)
  * Age: from 60 to 90 years old
  * Native language: French
  * Progressive deterioration of memory reported by patient or caregiver for more than 6 months
  * Profile at RL /RI 16: no significant improvement with indexing
  * Episodic memory disorder isolated or associated with other cognitive disorders
  * MRI: Atrophy of the median temporal lobe
  * Affiliation to a social security or to another social protection
  * Signature of informed consent

    • Healthy subjects
  * Healthy subject included in the BioHD protocol
  * MMS ≥ 26
  * Age from 18 to 90 years old
  * Native language: French
  * Affiliation to a social security or to another social protection
  * Signature of informed consent

Exclusion Criteria:

* Huntington's disease gene carriers

  * Intellectual deterioration preventing understanding of the protocol
  * Other dementia than Huntington's disease
  * Patient living alone at home
  * Major depression
  * Patient under legal protection
  * Patient deprived of liberty
  * Pregnant or breastfeeding woman, situation known to the investigator
  * Inability to handle an electronic tablet
* Patients with Alzheimer's disease

  * Intellectual deterioration preventing understanding of the protocol
  * Patient living alone at home
  * Sudden onset of memory impairment
  * Early onset of the following symptoms: difficulty in walking, convulsions, changes in behavior
  * Focal neurological characteristics including hemiparesis, sensory loss, visual field deficit
  * Early extrapyramidal sign
  * Other dementia than Alzheimer's disease
  * Major depression
  * Cerebrovascular disease
  * Toxic, metabolic or infectious anomaly
  * Patient under legal protection
  * Patient deprived of liberty
  * Pregnant or breastfeeding woman, situation known to the investigator
  * Inability to handle an electronic tablet
* Healthy subjects

  * Intellectual deterioration preventing understanding of the protocol
  * Known neurological or psychiatric illness
  * Patient under legal protection
  * Subject deprived of liberty
  * Pregnant or breastfeeding woman, situation known to the investigator
  * Inability to handle an electronic tablet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Ability to discriminate durations | 25 months and 10 days
  Ability to discriminate durations of a few seconds and durations of the order of minutes

SECONDARY OUTCOMES:
Risks's prediction of temporal disorientation. | 26 months
  Analysis of the answers (true/false) to the questionnaire assessing temporal orientation in daily life
Identification of neural correlations with temporal perception tests | 27 months
  Brain magnetic resonance imaging analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Catherine BACHOUD-LEVI, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - Hôpital Henri Mondor, Créteil, France